CLINICAL TRIAL: NCT02582216
Title: 3D Augmented Reality Mirror Visual Feedback Therapy Applied to the Treatment of Persistent, Unilateral Upper Extremity Neuropathic Pain: A Preliminary Study
Brief Title: 3D Augmented Reality Mirror Visual Feedback Applied to the Treatment of Unilateral Upper Extremity Neuropathic Pain.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Kine-001
Record Dates: First submitted 2015-10-01; First posted 2015-10-21 (Estimated); Results first posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Neuralgia
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label (Experimental): 3D augmented reality
  Interventions: Device: 3D augmented reality

INTERVENTIONS:
Device: 3D augmented reality — Each treatment period included a 3DARS (3D augmented reality system)training session.All 3DARS training sessions were performed in the same quiet room under the supervision of the same single investigator.The 3DARS training session protocol included two virtual training procedures. The first virtual training procedure consisted of applying a vertical virtual mirror to the display screen, where the non-affected side of the patient's body (such as the right) was symmetrically duplicated by a vertical axis on the affected side (such as the left).The second virtual training procedure consisted of flipping the 3D image horizontally along a vertical axis. This allowed patients to observe the reflection of their non-affected upper extremity as if it was the affected one.

SUMMARY:
This study has two objectives. First, to introduce a new virtual reality method that incorporates the mechanisms used in mirror visual feedback through a three-dimensional (3D) augmented virtual reality system. Second, to evaluate the efficiency of this new method on a convenience sample of patients presenting with unresolved neuropathic pain (CRPS, PLP, plexopathy, stroke) who were not responding adequately to both pharmaceutical management and traditional mirror therapy.

DETAILED DESCRIPTION:
Each patient receives 5 treatment periods over a total period of 1 week, where each treatment period lasts a total of 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Neuropathic pain in the unilateral upper extremity scored by DN4 questionnaire
* At least 3 months symptom duration following injury
* Minimum pain of 40 on a visual analogue scale (VAS);
* A drug treatment regimen that was stable for at least 2 weeks.
* Subjects were allowed to participate if they presented with any of the following: (1) A CRPS diagnosis, in accordance with the International Association for the Study of Pain criteria, Phantom Limb Pain (PLP), or spinal cord injury or plexopathy; and (2) an history of being treated before by conventional mirror therapy but, in their case, the mirror therapy failed.

Exclusion Criteria:

* Bilateral injury,
* Patients with epilepsy
* Side effects known to 3D (such as nausea, cephalalgia)
* Cognitive disorder
* Poor knowledge of the French language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open Label
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 22

OUTCOME MEASURES:

1. Primary Outcome: Pain on the Visual Analog Scale (VAS)
Description: Visual Analogic Scale assessed pain intensity before and after the intervention. Possible scores range from 0 (no pain) to 10 (worst possible pain)
Time Frame: baseline and week
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open Label: each patients received 5 3D augmented reality over a period of 5 days. Each treatment lasted a total of 20 minutes
Arm/Group | Open Label
Number analyzed (Participants) | 22
units on a scale
  vas baseline | 6.4 (2.3)
  vas after 1 week | 4.0 (2.4)

2. Secondary Outcome: Neuropathic Pain Assessed With DN4 Questionnaire
Description: DN4 (Douleur Neuropathique en 4 Questions) is a screening tool for neuropathic pain consisting of interview questions (DN4-interview) and physical tests.
  When the practitioner suspects neuropathic pain, the DN4 questionnaire is useful as a diagnostic tool.
  This questionnaire is divided into 4 questions representing 10 check items:
  * The practitioner questions the patient himself and completes the questionnaire
  * For each item, he must provide a "yes" or "no" answer
  * At the end of the questionnaire, the practitioner counts the responses, 1 for each "Yes" and 0 for each "no".
  * The sum obtained gives the Patient Score, noted out of 10.
  If the patient's score is 4/10 or more, the test is positive (sensitivity at 82.9%; specificity at 89.9%)
  Dn4 questionnaire were completed before and 24 hour after the last session
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open Label: Each patient received a 3D augmented reality
Arm/Group | Open Label
Number analyzed (Participants) | 22
units on a scale
  before | 6.5 (2.3)
  24H after the last treatment | 5.5 (2.3)

3. Other Pre Specified Outcome: Questionnaire de Saint-Antoine
Description: French adaptation of Melzack's MC Gill Pain Questionnaire (MPQ). It is a questionnaire of 61 qualifying words divided into 17 subclasses: 9 sensory, 7 emotional, 1 evaluative. The patient is asked to select the adjectives and then rate them from 0 (not at all) to 4 (extremely). This self-assessment scale allows clinical practice to specify the participation of the sensory and the emotional in pain intensity.
  self-questionnaire scoring the sensory and emotional qualities of the pain
Time Frame: 1 week
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Virtual training activities were terminated if patients complained about the development of headache or nausea, which are the most common side effects provoked by the use of stereovision systems similar to the 3DARS system. These symptoms were not present in this population.
Groups:
- Open Label: patients received a 3D augmented reality treatment
Arm/Group | Open Label
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No